CLINICAL TRIAL: NCT02267655
Title: An Exploratory, 3-Part, Clinical Study to Assess the Effect of Pulsed, Inhaled Nitric Oxide (iNO) on Functional Pulmonary Imaging Parameters in Subjects With World Health Organization (WHO) Group 3 Pulmonary Hypertension (PH) Associated With Chronic Obstructive Pulmonary Disease (COPD) on Long-Term Oxygen Therapy (LTOT) (Part 1) and in Subjects With WHO Group 3 PH Associated With Idiopathic Pulmonary Fibrosis (IPF) on LTOT (Part 2 and Part 3)
Brief Title: 3 Part Study to Assess Inhaled Nitric Oxide on Functional Pulmonary Imaging in Subj. Pulmonary Hypertension Associated w/ COPD and IPF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bellerophon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IK-7002-COPD-006
Record Dates: First submitted 2014-10-07; First posted 2014-10-17 (Estimated); Last update posted 2023-02-21 (Actual); Status verified 2017-08

CONDITIONS: Pulmonary Hypertension; Chronic Obstructive Pulmonary Disease; Idiopathic Pulmonary Fibrosis
Keywords: Inhaled Nitric Oxide (iNO); Pulmonary Hypertension (PH); Chronic Obstructive Pulmonary Disease (COPD); Long Term Oxygen Therapy (LTOT); Idiopathic Pulmonary Fibrosis (IPF)
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Disease, Chronic Obstructive; Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- inhaled Nitric Oxide 30 mcg/kg IBW/hr (Active Comparator): 30 mcg/kg IBW/hr of inhaled Nitric Oxide Part 1
  Interventions: Drug: inhaled Nitric Oxide - 30 mcg/kg IBW/hr
- inhaled nitric oxide 75 mcg/kg IBW/hr (Active Comparator): Part 2: 75mcg/Kg IBW/hr
  Interventions: Drug: inhaled nitric oxide 75 mcg/kg IBW/hr
- inhaled Nitric Oxide 5,10,15 mcg/Kg IBW/hr (Active Comparator): Part 3a: Dose tritration 5, 10 and 15 mcg/Kg IBW/hr Part 3b: continuing on dose determined by PI in 3a for 4 weeks
  Interventions: Drug: inhaled Nitric Oxide 5,10,15 mcg/Kg IBW/hr
- Placebo (Placebo Comparator): Placebo for 75 mcg/kg IBW/hr
  Interventions: Drug: inhaled nitric oxide 75 mcg/kg IBW/hr

INTERVENTIONS:
Drug: inhaled Nitric Oxide - 30 mcg/kg IBW/hr — inhaled Nitric Oxide in 30 mcg/kg IBW/hr doses Part 1
  Other Names: inhaled NO; inhaled Nitric Oxide; iNO
  Arms: inhaled Nitric Oxide 30 mcg/kg IBW/hr
Drug: inhaled Nitric Oxide 5,10,15 mcg/Kg IBW/hr — inhaled inhaled Nitric Oxide 5,10,15 mcg/Kg IBW/hr dose titration
  Other Names: inhaled NO; inhaled Nitric Oxide; iNO
  Arms: inhaled Nitric Oxide 5,10,15 mcg/Kg IBW/hr
Drug: inhaled nitric oxide 75 mcg/kg IBW/hr — inhaled nitric oxide 75 mcg/kg IBW/hr -Part 2b
  Other Names: iNO
  Arms: Placebo; inhaled nitric oxide 75 mcg/kg IBW/hr

SUMMARY:
The objective of this exploratory study is to examine the utility of high resolution computed tomography (HRCT) to measure changes in functional pulmonary imaging parameters as a function of short term a) iNO administration and b) nitric oxide (NO) cylinder concentration using the investigational medical device INOpulse® DS-C in subjects with WHO Group 3 PH associated with COPD on LTOT (Part 1) and in Subjects with WHO Group 3 PH associated with Idiopathic Pulmonary Fibrosis (IPF) on LTOT (Part 2 and Part 3)

DETAILED DESCRIPTION:
This is an exploratory, two-part, clinical study to evaluate the utility of HRCT to measure the pharmacodynamic effects of short term, pulsed administration of iNO using the combination product, inhaled nitric oxide/INOpulse in subjects with PH associated with COPD on LTOT. The utility of HRCT to characterize the effect of iNO on pulmonary imaging parameters as a function of a) short term inhaled iNO administration and b) NO cylinder concentration will be studied. In this study, pulmonary hypertension (PH) is defined as a tricuspid regurgitation velocity (TRV) ≥ 2.9 meters/second (m/s) or sPAP ≥ 38 mmHg by 2-D echocardiogram with Doppler or a mean pulmonary arterial pressure (mPAP) ≥ 25 mmHg by right heart catheterization.

Eleven subjects will be enrolled; the first 6 subjects enrolled will be assigned to Part 1, the next 2 subjects enrolled will be assigned to Part 2. After Part 1 has been completed and the results reviewed by the Sponsor, the next 4 subjects will be enrolled in Part 2. The Next three subjects will be participating in Part 3.

In Part 1, six (6) subjects with adequate kidney function will be randomized to receive the 30 mcg/kg IBW/hr doses of iNO using a cylinder concentration of 4880 ppm (6.0 mg/L).

The 2 subjects enrolled in Part 2a will be randomly assigned to 1 of 2 sequences (2 subjects/sequence) to receive iNO utilizing NO cylinder concentration (4880 ppm) at a dose of 75 mcg/kg IBW/hr or Placebo set at a dose of 75 mcg/kg IBW/hr . The 2 patients from Part 2a will enter Part 2b. During Part 2b patients will receive iNO utilizing NO cylinder concentration (4880 ppm) at a dose of 75 mcg/kg IBW/hr (INOpulse® setting of 75 mcg/kg IBW/hr) for 4 weeks for at least 12 hours/day.

The 3 subjects enrolled in Part 3a and 3b. Part 3a is dose titration visit, Part 3 is 4 weeks of treatment at dose identified in Paret 3a at the discretion of the Investigator. Part 3a: subjects will receive three different doses of iNO utilizing NO cylinder concentration of (4880ppm) at a dose of 5, 10 and 15 mcg/kg IBW/hr.

The 3 patients from Part 3a will enter Part 3b and will be administered open label iNO for 4 weeks/at least 12 hrs/day at the dose determined by the Investigator in Part 3a.

Subjects will be replaced if they are unable to complete all treatment visits or of evaluable HRCT data cannot be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following inclusion criteria to be enrolled and eligible to participate in the study:

  1. A confirmed diagnosis of COPD by the Global initiative for chronic Obstructive Lung Disease (GOLD) criteria
  2. Pulmonary hypertension determined by one of the following within the past 12 months:

     1. A right heart catheterization (not obtained within ± 7 days of an exacerbation) with an mPAP ≥ 25 mmHg, or
     2. An echocardiogram (not obtained within ± 7 days of an exacerbation) with a TRV ≥ 2.9 m/s or sPAP ≥ 38 mmHg (Note: a subject with an acceptable mPAP ≥ 25 mmHg determined by right heart catheterization will meet this inclusion criteria even with a TRV < 2.9 m/s)
  3. Current or former smokers with at least 10 pack-years of tobacco cigarette smoking before study entry
  4. Age ≥ 40 years, ≤ 80 years
  5. A post-bronchodilatory FEV1/FVC < 0.7 and a FEV1 < 60% predicted (values obtained within 6 months prior to screening can be used unless obtained within ± 7 days of an exacerbation; otherwise, the test must be performed during screening)
  6. Receiving LTOT for ≥ 3 months and ≥ 10 hours per day as determined by history
  7. Females of childbearing potential must have a negative pre-treatment urine pregnancy test
  8. Signed informed consent prior to the initiation of any study mandated procedures or assessments

Exclusion Criteria:

* Subjects who meet any of the following criteria are not eligible for enrollment:

  1. A diagnosis of asthma or other non-COPD respiratory disease, in the opinion of the Investigator
  2. Lack of patency of nares upon physical examination
  3. Experienced during the last month an exacerbation requiring:

     1. start of or increase in systemic oral corticosteroid therapy and/or
     2. hospitalization
  4. Left ventricular dysfunction as measured by:

     1. Screening echocardiographic evidence of left ventricular systolic dysfunction (left ventricular ejection fraction [LVEF] < 40%), or
     2. Screening echocardiographic evidence of left ventricular diastolic dysfunction

        > moderate (i.e., > Grade 2), or
     3. Any history of pulmonary capillary wedge pressure (PCWP), left atrial pressure (LAP) or left ventricular end diastolic pressure (LVEDP) > 18 mmHg as measured during cardiac catheterization within the past 6 months unless documented to have resolved by a subsequent cardiac catheterization
  5. Renal impairment (i.e., an estimated GFRMDRD < 60 ml/min/1.73 m2) or history of renal failure using the equation (Levey et al., 2007):

     estimated GFRMDRD = 175×Scr -1.154×Age-0.203 ×1.212 (if black) ×0.742 (if female)

     where Scr = Standardized serum creatinine
  6. Known allergy to contrast media.
  7. Clinically significant valvular heart disease that may contribute to PH, including mild or greater aortic valvular disease (aortic stenosis or regurgitation) and/or moderate or greater mitral valve disease (mitral stenosis or regurgitation), or status post mitral valve replacement
  8. Use within 30 days of screening or current use of approved PH medications such as sildenafil or bosentan (use of Cialis® or Viagra® for erectile dysfunction is permitted)
  9. Use of investigational drugs or devices within 30 days prior to enrollment into the study
  10. Any underlying medical or psychiatric condition that, in the opinion of the Investigator, makes the subject an unsuitable candidate for the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-05; Primary Completion 2017-06 (Actual); Study Completion 2017-06-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline in lobar blood volume at total lung capacity (TLC) after dosing with pulsed iNO as measured by HRCT | up to 4 weeks
  Part 1: baseline to end of treatment (1 day)
  Part 2: baseline to end of treatment (treatment visit B will occur at least 5 days and not more than 30 days after treatment visit A)

SECONDARY OUTCOMES:
Changes in baseline measured by HRCT after dosing with pulsed iNO in Blood vessel % and density on lobar level | up to 4 weeks
  Changes in baseline measured by HRCT after dosing with pulsed iNO in Blood vessel % and density on lobar level
Changes in baseline measured by HRCT after dosing with pulsed iNO in Total lung volume at TLC | up to 4 weeks
  Changes in baseline measured by HRCT after dosing with pulsed iNO in Total lung volume at TLC
Changes in baseline measured by HRCT after dosing with pulsed iNO in Lobar volumes at TLC | up to 4 weeks
  Changes in baseline measured by HRCT after dosing with pulsed iNO in Lobar volumes at TLC
Changes in baseline measured by HRCT after dosing with pulsed iNO in Internal airflow distribution based on lobar expansion | up to 4 weeks
  Changes in baseline measured by HRCT after dosing with pulsed iNO in Internal airflow distribution based on lobar expansion
Changes in baseline measured by HRCT after dosing with pulsed iNO in Airway volume down to generation 8-10 at TLC | up to 4 weeks
  Changes in baseline measured by HRCT after dosing with pulsed iNO in Airway volume down to generation 8-10 at TLC
Changes in baseline measured by HRCT after dosing with pulsed iNO in Computational Fluid Dynamics (CFD)-based resistance on lobar level | up to 4 weeks
  Changes in baseline measured by HRCT after dosing with pulsed iNO in Computational Fluid Dynamics (CFD)-based resistance on lobar level
Changes in baseline measured by HRCT after dosing with pulsed iNO in Ventilation/perfusion (V/Q) matching | up to 4 weeks
  Changes in baseline measured by HRCT after dosing with pulsed iNO in Ventilation/perfusion (V/Q) matching

CONTACTS AND LOCATIONS:
Overall Officials: Ashika Ahmed, Study Director — Bellerophon Therapeutics
Locations (1):
- Antwerp University Hospital, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No